CLINICAL TRIAL: NCT02069964
Title: A Prospective Longitudinal Cohort Study Looking at the Difference in Carotid Intima-medial Thickness Between Irradiated and Unirradiated Carotid Arteries in Patients With Head and Neck Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Royal Brompton and Harefield NHS Foundation Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: CCR 3688
Record Dates: First submitted 2014-02-18; First posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Head and Neck Tumours

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prospective hemi-neck RT

SUMMARY:
Some patients with head and neck cancer or benign tumours of the head and neck receive radiotherapy to their neck as part of their treatment. The large arteries in the neck, the carotid arteries, are often included in the area being treated with radiotherapy. There is some evidence to show that radiotherapy to these blood vessels can result in thickening and furring of the artery walls some years after treatment. This thickening may then result in stiffening and narrowing of the artery.

Current research is now aimed towards detecting radiotherapy-related changes to the carotid arteries at an earlier stage and towards using new radiotherapy techniques to avoid treating these blood vessels if possible. The question of whether or not the use of preventive medicines like aspirin and cholesterol-lowering tablets helps to reverse this process is currently unanswered.

The aim of this study is to compare the thickness (intima-medial thickness) of the carotid artery wall over time (a period of 5 years) following radiotherapy to the thickness in carotid arteries that have not received radiotherapy. There are many other causes for thickening of arteries (such as high blood pressure, high cholesterol levels and diabetes) and these may affect the ability to measure the effect of radiotherapy change to the artery wall. In order to address this, it is ideal to look at this process in patients who are having only one side of the neck treated and use the other side as a comparison. The study will also be investigating for earlier signs of radiotherapy-related changes, such as stiffening of the artery wall, inflammation in the artery wall (a very early sign of radiotherapy-related change) and some markers in the blood that may indicate that this process is taking place.

The null hypotheses of this study are:

* In irradiated carotid arteries, mean intimal-medial thickness at one year following radiotherapy will be the same as in unirradiated arteries.
* The incidence of carotid artery stenosis will be the same in irradiated and unirradiated carotid arteries
* Arterial wall strain at one year following radiotherapy will be the same in irradiated and unirradiated carotid arteries.
* Microbubble ultrasound will not be able to detect Inflammation in the carotid arteries during radiotherapy as an early marker of atherosclerosis; microbubble ultrasound will not demonstrate at what dose of radiotherapy inflammation begins.
* Serum biomarker levels will not increase over time from baseline after radiotherapy and won't correlate to IMT and arterial strain.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older
* Histologically confirmed cancer or benign tumours of the head and neck area requiring ≥ 50Gy to one side of the neck (conventional or intensity modulated RT)
* Prior or subsequent neck dissection allowed (irradiated and/or unirradiated side)
* Be able to provide written informed consent

Exclusion Criteria:

* Patients with bulky nodal neck disease that may interfere with acquisition of ultrasound images
* Patients with a prior history of carotid endarterectomy or carotid angioplasty and stenting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with histologically confirmed canceror benign tumours of the head and neck area requiring hemi-neck radiotherapy to ≥ 50Gy
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
The difference in mean carotid IMT at one year after radiotherapy between irradiated and unirradiated carotid arteries. | 1 year
  Measured at baseline and 12 months after radiotherapy

SECONDARY OUTCOMES:
The difference in mean carotid IMT at 2 and 5 years after radiotherapy between irradiated and unirradiated carotid arteries. | 2 and 5 years
  Measured at baseline, weekly during radiotherapy, 3 and 6 months after radiotherapy, then annually to 5 years
The incidence of carotid artery stenosis in irradiated carotid arteries compared to unirradiated carotid arteries. | 5 years
  Measured up to 5 years after radiotherapy
The difference in carotid arterial wall strain following radiotherapy between irradiated and unirradiated carotid arteries. | 5 years
  Measured at baseline, weekly during radiotherapy, 3 and 6 months after radiotherapy, then annually to 5 years
The difference in arterial wall inflammation between irradiated and unirradiated carotid arteries and dose-related effects | 5 years
  Measured at baseline, weekly during radiotherapy, 3 and 6 months after radiotherapy, then annually to 5 years
The effect of risk-modifying therapy (anti-hypertensives, anti-diabetic medication, HMGCoA reductase inhibitors, smoking cessation) on irradiated and unirradiated carotid arteries. | 5 years
  Measured at baseline, 3 and 6 months after radiotherapy, then annually to 5 years
The change in mean serum biomarker levels after radiotherapy. | 1 year
  Baseline, week 6 after radiotherapy, then 3-, 6-, and 12 months after radiotherapy
The proportion of patients who develop stroke or TIA. | 5 years
  The proportion of patients who develop stroke or TIA during the trial period

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Nutting, PhD, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital, London, United Kingdom